CLINICAL TRIAL: NCT00401284
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Hypnotic Efficacy of EVT 201 in Elderly Patient With Daytime Sleepiness
Brief Title: Efficacy Study of EVT 201 in the Treatment of Elderly Patients With Daytime Sleepiness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evotec Neurosciences GmbH (Industry)
Organization: Evotec International GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — EVT 201

INTERVENTIONS:
Drug: EVT 201

SUMMARY:
The purpose of this study is to determine whether a compound known as EVT 201 is effective in treating elderly patients diagnosed with primary insomnia who also have moderate daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia according to DSM-IV
* Over the last three months for at least 5 nights per week, must have a normal bedtime of between 9 pm and 1 am and a time in bed of at least 7 hours
* A history of sleepiness, tiredness or unintentional napping during the daytime attributed to to poor sleep at night
* Able to attend the Sleep Center for five nights (two consecutive nights on two occasions and one night on one occasion)over a five week period
* Willing and able to complete a sleep diary and questionnaires

Exclusion Criteria:

* Clinically significant or unstable medical condition that may interfere with sleep
* Major psychiatric disorders (other than insomnia) such as depression, schizophrenia, bipolar disorder
* History of myocardial infarction, cardiac failure or clinically significant dysrhythmias in the previous 2 years or clinically significant ECG abnormalities at screening
* History of substance abuse
* Disorders that interfere with drug pharmacokinetics
* History of cancer, except basal cell carcinoma
* Use of hypnotics, anxiolytics, antidepressants, anticonvulsants, over-the-counter sleep aids, histamine-1 receptor antagonists (except for loratadine and fexofenadine), beta-adrenergic blockers (except for atenolol), respiratory stimulants and decongestants, systemic steroids, narcotic analgesics, any other compound which might impact sleep-wake function, or medication used for the treatment of Parkinson's disease such as dopamine agonists and L-dopa (e.g., Sinemet, Madopar or Requip)
* Use of hypnotics within the 2 weeks preceding the Screening Period or within five half-lives of the medication, whichever is longer
* Consuming ≥ 350 mg per day of xanthine-containing food or beverages
* Smoking ≥ 10 cigarettes per day and/or unable to refrain from smoking without distress or discomfort for the duration of visits to the sleep laboratory (i.e.≥ 20 hours)
* Body mass index > 34 kg/m2;
* Performing night work or rotating shift work during the past month
* Traveling across > 3 time zones in the past 2 weeks
* Participation in another trial of an investigational product or device within the previous 30 days
* Known allergy or sensitivity to benzodiazepines

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2006-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Polysomnography derived Total Sleep Time averaged over nights 1, 6 and 7

SECONDARY OUTCOMES:
Mean Multiple Sleep Latency Test at Day 8
Mean Psychomotor Vigilance Task at Day 8
Mean Karolinska Sleepiness Scale at Day 8
Mean Rey Auditory Verbal Learning Test at Day 8
Mean Profile of Mood State at Day 8
Polysomnography derived variables averaged over nights 1, 6 and 7
Patient reported evaluations of sleep quality and quantity over nights 1 to 7
Benzodiazepine withdrawal questionnaire at baseline and follow-up
Safety including adverse events, ECGs, vital signs, routine laboratory tests throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: James K Walsh, PhD, Principal Investigator — St Luke's Hospital, Sleep Medicine and Research Center, Chesterfield, MI
Locations (22):
- United States (22):
  - PsyPharma Clinical Research Inc., Phoenix, Arizona
  - PsyPharma Clinical Research, Inc., Tucson, Arizona
  - Pacific Sleep Medicine Services Inc, Los Angeles, California
  - Pacific Sleep Medicine Services, San Diego, California
  - Miami Research Associates, Miami, Florida
  - OmniTrials, 11181 Health Park Blvd, Suite 3040, Naples, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Clinical Research Group of St Petersburg Inc., 2525 Pasadena Ave So, Suite S, St. Petersburg, Florida
  - The Sleep Disorders Center of Georgia, Peachtree Dunwoody Medical Center, 5505 Peachtree Dunwoody Road, Suite 548, Atlanta, Georgia
  - Sleep Disorders Center of Georgia - Gainesville, Gainesville, Georgia
  - Vince and Assocaites Clinical Research, Overland Park, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Center for Sleep Medicine, 101 Courtney Circle, Hattiesburg, Mississippi
  - Sleep Medicine and Research Center, 232 S. Woods Mill Road, Chesterfield (St Louis), Missouri
  - Clinilabs, Inc., 423 West 55th Street, 4th Floor, New York, New York
  - Duke Insomnia and Sleep Research, Duke South Hospital, Room 54242, Trent Drive, Durham, North Carolina
  - Community Research, Cincinnati, Ohio
  - Tri-State Sleep Disorders Center, 1275 East Kemper Road, Cincinnati, Ohio
  - Bradley Hospital Sleep Research Laboratory, 300 Duncan Drive, Providence, Rhode Island
  - Sleep Disorders Center, 1333 Taylor Street, Suite 5A, Columbia, South Carolina
  - Sleep Medicine Associates p.a., 5477 Glen Lakes Drive, Suite 125, Dallas, Texas
  - Baylor College of Medicine, VAMC-Sleep Laboratory, 2002 Holcombe Boulevard , Room 6C-344, Houston, Texas